CLINICAL TRIAL: NCT06545461
Title: Treating Metabolic Acidosis in Chronic Kidney Disease to Prevent Adverse Kidney and Cardiovascular Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-INTMED-97884
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases; Hypertension
Keywords: acidosis; albuminuria; diet
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Hypertension; Acidosis; Albuminuria | interventions — Fruit; Vegetables; Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: prospective, randomized parallel three-arm design
Masking Description: None (Open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fruits and vegetables (F+V) (Experimental): 36 participants with hypertension, eGFR 30-59 ml/min/m2, macroalbuminuria (albumin [mg] to creatinine [g] ratio > 200 mg/g) and PTCO2 >22 but <24 mM will receive a prescribed amount of F+Vs designed to reduce dietary acid intake by half. The chosen level of metabolic acidosis does not warrant alkali treatment by current guidelines with standard therapy, oral NaHCO3. Because macroalbuminuria places them at increased risk for worsening kidney function and development of CVD, they will receive oral enalapril (minimum 5 mg daily) and oral atorvastatin (minimum 10 mg daily). They will otherwise receive standard medical care and followed annually for 10 years.
  Interventions: Other: Fruits and Vegetables (F+V)
- NaHCO3 (HCO3) (Experimental): 36 participants with hypertension, eGFR 30-59 ml/min/m2, macroalbuminuria (albumin [mg] to creatinine [g] ratio > 200 mg/g) and PTCO2 >22 but <24 mM will receive sodium bicarbonate (NaHCO3) dosed to match the alkali intake of the F+V given to the F+V group. Because macroalbuminuria places them at increased risk for worsening of their kidney function and for development of CVD, they will receive oral enalapril (minimum 5 mg daily) and oral atorvastatin (minimum 10 mg daily). They will otherwise receive standard care and followed annually for 10 years.
  Interventions: Other: Sodium Bicarbonate (NaHCO3)
- Usual Care (UC) (Active Comparator): 36 participants with hypertension, eGFR 30-59 ml/min/m2, macroalbuminuria (albumin [mg] to creatinine [g] ratio > 200 mg/g) and PTCO2 >22 but <24 mM will receive no additional alkali (neither F+V or NaHCO3). The chosen level of metabolic acidosis does not warrant alkali treatment by current guidelines with standard therapy with oral NaHCO3. Because their macroalbuminuria places them at increased risk for worsening of their kidney function and for subsequent development of CVD, they will receive oral enalapril (minimum 5 mg daily) and oral atorvastatin (minimum 10 mg daily). They will otherwise receive standard care and followed annually for 10 years.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Fruits and Vegetables (F+V) — Participants will receive a prescribed amount of F+V designed to reduce their dietary acid intake by half. This typically amounts to 2-4 cups daily of F+V provided in weekly allotments. Amount provided will be that calculated for the participant multiplied times number of household members to assure participants eat the prescribed amount and do not share with household members.
  Arms: Fruits and vegetables (F+V)
Other: Sodium Bicarbonate (NaHCO3) — Participants will receive 0.3 mEq/kg bw/day NaHCO3 tablets to match the alkali provided by F+V given to F+V participants. This will be provided as 650 mg NaHCO3 tablets for an average of 4-5 tablets/day in two divided oral doses.
  Arms: NaHCO3 (HCO3)
Other: Usual Care — Participants will receive standard medical care but no additional alkali (F+V nor NaHCO3).
  Arms: Usual Care (UC)

SUMMARY:
Upon completion, this project will determine if treatment of metabolic acidosis in non-diabetic study participants with reduced kidney function (chronic kidney disease [CKD] stage 3) associated with high blood pressure (hypertension) and macroalbuminuria, the latter indicating pronounced kidney injury, using either base-producing fruits and vegetables (F+V) or standard therapy for treatment of metabolic acidosis with the medication sodium bicarbonate (NaHCO3) 1) slows progression of CKD toward end-stage renal disease [ESRD]; 2) improves indices of cardiovascular disease (CVD) risk; and 3) better preserves plasma acid-base parameters. These studies are designed to compare the differential effects of treating the metabolic acidosis of CKD with F+Vs or NaHCO3 on kidney outcomes, including progression to ESRD, on indices of CVD risk and on plasma acid-base parameters.

DETAILED DESCRIPTION:
The long-term objective of this study is to determine if treatment of metabolic acidosis in study participants with chronic kidney disease (CKD), reduced estimated glomerular filtration rate (eGFR), and very high levels of urine albumin excretion (macroalbuminuria) reduces risk for further eGFR decline and/or for subsequent development of cardiovascular disease (CVD). The specific aims of this study are to determine if metabolic acidosis treatment with either base-producing fruits and vegetables (F+V) in amounts calculated to reduce participant dietary acid content by half, or sodium bicarbonate (NaHCO3, 0.3 mEq/kg body weight, an amount designed to match the alkali content of provided F+V) in participants with stage 3 CKD (eGFR 30 to 59 ml/min/1.73 m2) compared with Usual Care 1) slows CKD progression; 2) improves indices of cardiovascular risk; and 3) better preserves plasma acid-base parameters. Despite blood pressure control with "kidney protective" drugs like angiotensin converting enzyme (ACE) inhibitors, many patients with CKD and reduced eGFR have progressive eGFR decline toward end-stage renal disease (ESRD) with need for dialysis or kidney transplant to maintain life. They also have increased risk to die of CVD. Studies from our laboratory and those of other investigators support that treatment of metabolic acidosis slows GFR decline in animal models of CKD. Many patients with CKD stage 3 have metabolic acidosis that might exacerbate eGFR decline and its treatment might slow or stop it. This study will recruit participants with hypertension-associated CKD stage 3 (eGFR 30-59 ml/min/1.73 m2) without diabetes to avoid contribution of diabetes to eGFR decline. They will have macroalbuminuria (urine albumin [mg]-to-creatinine [g] ratio > 200 mg/g) that increases their CKD progression risk to optimize the chance to see benefits of metabolic acidosis treatment. They will have plasma total CO2 (PTCO2) < 24 but > 22 millimolar (mM) to recruit participants with metabolic acidosis that is not severe enough to warrant treatment by current guidelines (with oral NaHCO3) to ethically randomize participants to received non-recommended treatment for metabolic acidosis (F+V) or no treatment (Usual Care). Participants whose PTCO2 decreases to 22 mM or below during follow up will be treated with oral NaHCO3 tablets with the goal to maintain their PTCO2 > 22 mM. All will undergo blood pressure control to target systolic blood pressure < 130 mm Hg (millimeters of mercury) with regimens including ACE inhibition and will receive atorvastatin because their macroalbuminuria puts them at increase CVD risk. At study entry and yearly for 10 years, all participants will have 10 ml of blood drawn from an antecubital vein for measurement of the negative log of free hydrogen ion concentration (pH), partial pressure of carbon dioxide gas (PCO2), PTCO2, creatinine, LDL cholesterol, HDL cholesterol, Lp(a) cholesterol, sodium, potassium, and chloride. They will have 20 ml of urine collected for measurement of creatinine, albumin, N-acetyl-D-glucosaminidase, angiotensinogen, and isoprostane 8-isoprostaglandin F2 alpha. They will also have an 8-hour urine collection at a Texas Tech University Health Sciences Center (TTUHSC) clinic at baseline, 3 years, 5 years, and 10 years for PTCO2, pH, ammonium, titratable acidity, creatinine, sodium, and potassium after fasting after midnight. The course of plasma and urine parameters over the 10 years of follow up in those randomized to F+V or NaHCO3 compared to Usual Care will help determine the effect(s) treatment of metabolic acidosis on CKD progression (change in urine indices of kidney injury and eGFR), indices of CVD risk (change in LDL, HDL, and Lp(a) cholesterol), and on participant acid-base status (serum acid-base parameters [pH, PCO2, bicarbonate concentration [HCO3], and PTCO2). These studies will also determine differences in metabolic acidosis treatment with F+V vs. NaHCO3. We hypothesize that metabolic acidosis treatment with F+V or NaHCO3 will 1) slow CKD progression indicated by lower urine kidney injury indices and slower eGFR decline; 2) improve indices of cardiovascular risk indicated by lower LDL, lower Lp(a), and higher HDL cholesterol; and 3) improve plasma acid-base status indicated by higher PTCO2. Excretion of urine acid-base parameters will help determine effects of these treatments on urine acid excretion. Blood pH and PCO2 will be measured using the Immediate Response Mobile Analysis (IRMA) blood analysis system and blood and urine concentrations of albumin and creatinine will be measured with standard techniques. Blood and urine PTCO2 will be measured as done previously with fluorimetry in the PI's laboratory. Urine ammonium, titratable acidity, N-Acetyl-beta-D-glucosaminidase, angiotensinogen, and isoprostane 8-isoprostaglandin F2 alpha will be measured as done previously in the laboratory of the Co-PI.

ELIGIBILITY:
Inclusion Criteria:

1. Non-malignant high blood pressure or hypertension
2. 18-70 yrs old
3. urine albumin-to-creatine ratio > 200 mg/g creatinine
4. estimated glomerular filtration rate (eGFR) 30 to 59 ml/min/1.73 m2
5. Plasma total CO2 (PTCO2) > 22 but < 24 mmol/l
6. able to tolerate angiotensin converting enzyme [ACE] inhibition drug therapy because guidelines recommend it for patients with albuminuric CKD
7. non-smoking
8. greater than or equal to 2 primary care visits in the preceding year, indicating compliance
9. Able to provide informed consent.

Exclusion Criteria:

1. Malignant hypertension or history thereof
2. primary kidney disease or findings consistent thereof such as > 3 red blood cells per high powered field of urine or urine cellular casts
3. history of diabetes or fasting glucose greater than or equal to 110/mg/dl
4. history of hematologic disorders, malignancies, chronic infections, current pregnancy, history or clinical evidence of CVD
5. peripheral edema or diagnosis associated with edema such as heart/liver failure or nephrotic syndrome because of the sodium load that accompanies NaHCO3 therapy
6. baseline plasma potassium concentration > 4.6 mmol/l to reduce the risk for hyperkalemia in those participants randomized to F+Vs which increases dietary potassium intake
7. taking, or unable to stop taking, drugs other than ACE inhibitors that limit urine potassium excretion
8. Unable to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 1998-06-22 (Actual); Primary Completion 2006-10-25 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Difference in estimated glomerular filtration rate (eGFR) at follow up | eGFR will be measured at baseline and yearly for 10 years
  eGFR (ml/min/1.73 m2) will be calculated using measured serum creatinine and cystatin-C concentrations, age, sex, and whether or not of African American ethnicity using a standard accepted formula.
  eGFR will be compared among the three groups yearly up to 10 years follow up to assess chronic kidney disease (CKD) progression. Milestone assessments will be done at 3, 5, and 10 years. Higher eGFR indicates better-preserved kidney function. The investigators hypothesize that F+V or NaHCO3 will lead to better preserved (higher) eGFR.
Difference in the rate of eGFR change during follow up | eGFR rate of change will be measured at 3, 5, and 10 years
  The rate of eGFR change (ml/min/1.73 m2/year) will assess CKD progression. It will be calculated by dividing the net change in eGFR between the milestone year of follow up and baseline divided by the years of follow up. The investigators hypothesize that F+V or NaHCO3 will lead to a slower rate of eGFR change, indicative of slower CKD progression.
Difference in the net eGFR change during follow up | eGFR net change compared to baseline will be measured at 3, 5, and 10 years
  The net eGFR change (ml/min/1.73 m2) will assess CKD progression and will be calculated by subtracting the milestone value from the baseline value. The investigators hypothesize that dietary acid reduction will lead to a smaller net eGFR change, indicative of less CKD progression.
Difference in the number of participants who reach need for kidney replacement therapy (KRT) | Number of participants reaching KRT will be determined at years 3, 5, and 10 from baseline
  Differences in the number of participants who reach the need for KRT will be determined by comparing the number of participants among arms who reach the need for dialysis or kidney transplant; this is a measure of how well the interventions protect kidney health. The investigators hypothesize that the F+V or NaHCO3 arms will have fewer participants reaching KRT.
Difference in change in urine albumin excretion during follow up | UACR will be measured at baseline and yearly for 10 years
  CKD progression will be assessed by change in the urine albumin (mg)-to-creatinine (g) ratio (UACR) in a "spot" urine. An increased UACR is indicative of kidney injury and risk for subsequent decrease of kidney function with time. A decrease in UACR is indicative of reduced kidney injury and a lower risk for decreased kidney function with time. The investigators hypothesize that F+V or NaHCO3 will lead to a lower UACR.
  • UACR will be compared among the three groups as follows: Value at 3,5, and 10 years Net change compared to baseline value at 3, 5, and 10 years
Difference in change in urine N-acetyl-D -glucosaminidase (UNAG) excretion during follow up | UNAG will be measured at baseline and yearly for 10 years
  CKD progression will be assessed by change in the UNAG (Units)-to-creatinine (g) ratio in a "spot" urine. An increased UNAG/creatinine ratio is indicative of increased kidney injury. The investigators hypothesize that F+V or NaHCO3 will lead to a lower UNAG/creatinine.
  • UNAG/creatinine will be compared among the three groups as follows: Value at 3, 5, and 10 years Net change compared to baseline at 3, 5, and 10 years
Difference in change in urine angiotensinogen (UATG) excretion during follow up | UATG will be measured at baseline and yearly for 10 years
  CKD progression will be assessed by change in the UATG (ug)-to-creatinine (g) ratio in a "spot" urine. An increased UATG/creatinine ratio is an indirect measure of kidney levels of angiotensin II and is indicative of increased kidney injury. The investigators hypothesize that F+V or NaHCO3 will lead to a lower UATG/creatinine ratio.
  • UATG/creatinine will be compared among the three groups as follows: Value at 3, 5, and 10 years Net change compared to baseline at 3, 5, and 10 years

SECONDARY OUTCOMES:
Difference in change in serum LDL cholesterol level during follow up | Serum LDL cholesterol will be measured at baseline and yearly for 10 years
  Higher serum LDL cholesterol levels (mg/dl) are an indicator of increased cardiovascular disease (CVD) risk. The investigators hypothesize that F+V leads to lower LDL cholesterol than that done with either NaHCO3 or Usual Care.
  Comparisons among the three groups will be done as follows:
  1. level at 3, 5, and 10 years
  2. Net change compared to baseline at 3, 5, 10 years
Difference in change in serum HDL cholesterol level during follow up | Serum HDL cholesterol will be measured at baseline and yearly for 10 years
  Higher serum HDL cholesterol levels (mg/dl) are an indicator of decreased CVD risk. The investigators hypothesize that F+V leads to higher HDL cholesterol than that done with either NaHCO3 or Usual Care.
  Comparisons among the three groups will be done as follows:
  1. level at 3, 5, and 10 years
  2. Net change compared to baseline at 3, 5, and 10 years
Difference in change in serum Lp(a) cholesterol level during follow up | Serum Lp(a) cholesterol will be measured at baseline and yearly for 10 years
  Higher serum Lp(a) cholesterol levels (mg/dl) are an indicator of higher CVD risk. The investigators hypothesize that F+V leads to lower Lp(a) cholesterol than either NaHCO3 or Usual Care.
  Comparisons among the three groups will be done as follows:
  1. level at 3, 5, and 10 years
  2. Net change compared to baseline at 3, 5, and 10 years
Difference in change in urine isoprostane 8-isoprostaglandin F2α excretion follow up | Urine Isoprostane 8-isoprostaglandin F2α to creatinine ratio will be measured at baseline and yearly for 10 years.]
  Higher urine excretion of isoprostane 8-isoprostaglandin F2α (U8-iso) is an indicator of increased oxidative stress which contributes to increased CVD risk. It will be measured as 8-iso (ug)-to-creatinine (g) ratio in a "spot" urine. The investigators hypothesize that F+V or NaHCO3 lead to a lower urine 8-iso/creatinine ratio.
  Comparisons among the three groups will be done as follows:
  1. level at 3, 5, and 10 years
  2. Net change compared to baseline at 3, 5, and 10 years
Difference in change in plasma pH during follow up | Plasma pH will be measured at baseline and yearly for 10 years
  Plasma pH (pH is expressed numerically without units) will be measured with standard blood gas machine techniques. The investigators hypothesize that F+V or NaHCO3 will lead to higher values for plasma pH.
  Comparisons among the three groups will be as follows:
  * Levels at 3, 5, and 10 years
  * Net change compared to baseline at 3, 5, and 10 years
Difference in change in plasma partial pressure of carbon dioxide gas (PCO2) during follow up | Plasma PCO2 will be measured at baseline and yearly for 10 years
  Plasma PCO2 [millimeter (mm) mercury (Hg)], will be measured with standard blood gas machine techniques. The investigators hypothesize that F+V or NaHCO3 will lead to higher values for plasma PCO2.
  Comparisons among the three groups will be as follows:
  * Levels at 3, 5, and 10 years
  * Net change compared to baseline at 3, 5, and 10 years
Difference in change in plasma bicarbonate concentration (HCO3-]) during follow up | Serum [HCO3-] will be measured at baseline and yearly for 10 years
  Plasma [HCO3-] (mEq/l) will be calculated from measured values of plasma pH and plasma partial pressure of carbon dioxide gas (PCO2) with a conventional formula commonly used by clinical laboratories. The investigators hypothesize that F+V or NaHCO3 will lead to higher values for plasma [HCO3-].
  Comparisons among the three groups will be as follows:
  * Levels at 3, 5, and 10 years
  * Net change compared to baseline at 3, 5, and 10 years
Difference in change in plasma total CO2 (TCO2) during follow up | Plasma TCO2 will be measured at baseline and yearly for 10 years
  Plasma TCO2 [millimolar (mM)] will be measured by the PI as in previous studies using fluorimetry. This technique uses an enzymatic assay in which TCO2 reacts with phosphoenolpyruvate to form oxaloacetate, which is reduced to malate coupled with oxidation of nicotinamide adenine dinucleotide bound to hydrogen ion (NADH) to nicotinamide adenine dinucleotide without hydrogen ion (NAD+). NADH fluoresces but NAD+ does not, allowing for quantitation of TCO2 as reduced fluorescence. This technique is more reproducible than the conventional one of measuring CO2 gas released upon addition of a strong acid.
  Measuring changes in plasma TCO2 will help assess the effect(s) of dietary acid reduction among the three groups. The investigators hypothesize that F+V or NaHCO3 will lead to higher values for plasma TCO2.
  Comparisons among the three groups will be as follows:
  * Levels at 3, 5, and 10 years
  * Net change compared to baseline at 3, 5, and 10 years

IPD SHARING:
Plan to Share IPD: Yes
Upon request, will provide study data and analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 90 days and for 30 days
Access Criteria: Other medical science investigators